CLINICAL TRIAL: NCT00164814
Title: Is Visceral Hyperalgesia the Culprit of Noncardiac Chest Pian in Chinese? Part I: The Role of Visceral Hyperalgesia, Gastroesophageal Reflux Disease (GERD) and Esophageal Motility Disorder (EMD) in NCCP Patients
Brief Title: The Role of Visceral Hyperalgesia, Gastroesophageal Reflux Disease (GERD) and Esophageal Motility Disorder (EMD) in NCCP Patients
Status: Terminated | Type: Observational
Why Stopped: Funding ended
Sponsor: Chinese University of Hong Kong (Other)
Other Study IDs: NPA study
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Non-Cardiac Chest Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Noncardiac chest pain (NCCP) is a common clinical problem worldwide. In Hong Kong, it has been estimated that about 20% of patients with chest pain are misdiagnosed to have coronary heart disease. Despite its benign nature, this condition causes anxiety, impairs quality of life and consumes a substantial amount of healthcare resources. While acid reflux and motility disorder in the esophagus are often attributed as the cause of NCCP, visceral hyperalgesia of esophagus is now recognized to play a central role in the pathogenesis of this condition. This research project aims to evaluate the role of visceral hyperalgesia in Chinese patients with NCCP. NCCP patients will be evaluated for the prevalence of gastroesophageal reflux disease and esophageal motility disorder by endoscopy, manometry and pH study. The visceral sensory and pain thresholds of these patients will be compared with asymptomatic controls.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with monthly angina-like chest pain and negative coronary angiogram or scintigraphy
* Age between 18-70

Exclusion Criteria:

* Gastroesophageal reflux disease
* Psychiatric illness
* Cerebrovascular accident
* Active peptic ulceration
* Heart failure or cardiac bradyarrhythmia
* Epilepsy
* Pregnancy or lactating female
* Previous hypersensitivity to muscle relaxant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin CY WU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China